CLINICAL TRIAL: NCT03837210
Title: Comparative Anti Helicobacter Pylori Efficacy Assessment of Unani Formulation and Quintuple Regimen
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Syed Zahoor Ul Hassan Zaidi, Syed Zahoor Ul Hassan Zaidi, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zahoor11
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: H.Pylori Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Drug (Experimental): This group is treated with Herbal formulation.
  Interventions: Drug: Pylorin
- Control Drug (Active Comparator): This group is treated with Quintuple therapy
  Interventions: Drug: Pylorin

INTERVENTIONS:
Drug: Pylorin — Poly Herbal formulation
  Other Names: Poly Herbal formulation

SUMMARY:
Helicobacter pylori (H. pylori) is a bacterium its infection is regarded the most common medical condition associated with gastritis1 more over peptic ulcer disease2, gastric adenocarcinoma3 and lymphoma.4control of H pylori infection is thought to be the solution of public health problem.5,6 rate of infection is abating in developed world 7 , but this is slow and people health is challenged, to stop or decrease the new cases is complicated despite the fact that route of transmission are still unclear .8-10 The only option for reducing incidence and prevalence is that screening of masses followed by eradication therapy. A rough estimate propose about 50% of developing country population is affected from infection than the industrialized country. Infected individual may be asymptomatic or some time present with gastroduodenal disease. Prevalence of H pylori is different in developing countries where the adult prevalence reaches up to 80% and in children it is found before the age of 10 years.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a bacterium its infection is regarded the most common medical condition associated with gastritis1 more over peptic ulcer disease2, gastric adenocarcinoma3 and lymphoma.4control of H pylori infection is thought to be the solution of public health problem.5,6 rate of infection is abating in developed world 7 , but this is slow and people health is challenged, to stop or decrease the new cases is complicated despite the fact that route of transmission are still unclear .8-10 The only option for reducing incidence and prevalence is that screening of masses followed by eradication therapy. A rough estimate propose about 50% of developing country population is affected from infection than the industrialized country. Infected individual may be asymptomatic or some time present with gastroduodenal disease. Prevalence of H pylori is different in developing countries where the adult prevalence reaches up to 80% and in children it is found before the age of 10 years.

Aims and objectives

1. To establish and evaluate scientific and clinical evidence of herbal/eastern formulation and find out the clinical safety and efficacy.
2. To measure the clinical response of herbal formulation in the patients of H.Pylori.

Research Questions

1. has the Unani formulation better effects than quadruple regimen?

Hypothesis (H1): Unani has shown better clinical, effects than quadruple regimen.

Null Hypothesis (Ho): Quadruple regimen has shown superior clinical, response than Unani formulation.

Experimental approaches

To check this hypothesis independent variable to dependent variable and perplexing variables will apply by statistical analysis. In this study H. Pylori infection, quadruple regimen are independent variables while signs and symptoms, level of improvement are dependent variables.

ELIGIBILITY:
Inclusion Criteria:

1. The individuals suffering from H. pylori infection .
2. Individuals having no previous history of H. pylori infection treatment.
3. Individuals living in Karachi.
4. Individuals with no pathological finding on routine examination.
5. Individuals from either socioeconomic class including lower, middle and higher.
6. Both male and female individuals between 14 to 55 years of age
7. Subjects with informed written consent
8. Patients having no complications regarding other than GIT system.

Exclusion Criteria

The following were the reason for excluding the individuals from this trial:

1. Patient with simultaneous physical illness, for example renal dialysis and uncontrolled diabetes mellitus.
2. Individuals having stomach or intestinal surgical history were excluded.
3. Individuals with past record of any herbal or allopathic medication were excluded
4. Individuals with hyper sensitivity history of drug or adverse reaction to any of the study drugs .
5. Females with pregnancy were also excluded for the safety measures
6. Individuals with coma, meningitis, and encephalitis or head injury were also excluded.
7. Hospitalized individuals due to any serious diseases were excluded.
8. Individuals with known poor compliance and history of drug abuse were excluded.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Eradication of H. Pylori | 4 week duration
  Negative Stool antigen for H. pylori

CONTACTS AND LOCATIONS:
Overall Officials: Zahoor Zaidi, M.Phil, Principal Investigator — Hamdard University

IPD SHARING:
Plan to Share IPD: No